CLINICAL TRIAL: NCT04120532
Title: Effects of Health Education for Patients Received Minimally Invasive Lumbar Spinal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N201904001
Record Dates: First submitted 2019-10-06; First posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Low Back Pain; Lumbar Degenerative Disease
Keywords: rehabilitation; Lumbar degenerative disease; Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education group (Experimental)
  Interventions: Behavioral: Perioperative Rehabilitation
- Usual care group (No Intervention)

INTERVENTIONS:
Behavioral: Perioperative Rehabilitation — Physical therapist will be consulted one day before and after the operation (OP) day. On the day before the OP day, they focus on education, including how to get up from bed and stand up from a chair. Five rehabilitation exercises are also demonstrated: 1) ankle flexion and extension, 2) knee flexion and extension, 3) hip joint abduction and adduction, 4) hip joint flexion and extension, and 5) drawing-in maneuver. The participants will be required to repeat each component to confirm that they can do it correctly. Each exercise is suggested to be done 10 times per day following MI-TLIF, and the number will be recorded 3 days (pre-OP day, post-OP day, and post-OP day 2).
  Arms: Education group

SUMMARY:
Lumbar degenerative disease surgery has been a routine clinical operation, and has good treatment effects. Although the patient's neurological symptoms improve after surgery, many patients still have postoperative muscle soreness. The postoperative rehabilitation intervention for the patients receiving traditional lumbar surgery has been confirmed to effectively improve pain and disability. However, in recent years, minimally invasive lumbar spinal surgery has gradually replaced traditional surgery, postoperative pain has been greatly reduced. Therefore, patients have the opportunity to receive early intervention in rehabilitation, but there is no standardization process for rehabilitation of minimally invasive lumbar spine surgery. Therefore, this study aims to establish a health education program for patients receiving minimally invasive lumbar spinal surgery, and conduct clinical trials to test its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 and 90 years old.
* Low back pain has been persisting at least 3 months.
* Clinical degeneration diagnosis supports the need of MI-TLIF.
* Able to understand Chinese.

Exclusion Criteria:

* Emergency surgery.
* Unstable vital sign.
* Any psychological, neurological, orthopedics, cardiopulmonary, and cancer history.
* Had spinal surgery before.
* Pregnancy.

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-04-25 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Change of Oswestry Disability Index | The day before operation day, and 1, 3, 6 months after surgery
  This scale evaluates subject's physical function. The range is 0 to 1. Higher values represent a better outcome.
Change of Visual Analogue Scale | The day before operation day, and 1, 3, 6 months after surgery
  This scale evaluates subject's pain intensity. "0" indicates no pain and "10" indicates the worst possible pain.
Change of Short Form 12 version 2 | The day before operation day, and 1, 3, 6 months after surgery
  This scale evaluates subject's health-related quality of life. We will record the subscales: physical component summary (PCS) and mental component summary (MCS). Higher values represent a better outcome.
Change of Functional reach test | The day before operation day, and 1, 3, 6 months after surgery
  It is a dynamic measure of balance. A 100 cm yardstick will be horizontally set on the wall with the acromion height. The patient will be asked to make a fit and reach forward as far as possible without moving his/her feet. It will be measured twice and the better outcome will be recorded.
Change of 30-second Chair Rise | The day before operation day, and 1, 3, 6 months after surgery
  It is used to evaluate the lower limb function and strength relating to the daily activities. The patient starts with a sitting position, and need to repeat stand-to-sit movements. He/She will be encouraged to move safely as soon as possible in 30 minutes. Higher number indicates better function.
Change of Timed Up and Go test | The day before operation day, and 1, 3, 6 months after surgery
  It was developed to measure subjects' balance and mobility. The patient starts with a sitting position, stands up, walks a 3-meter distance, turns, walks back, and sits down. He/She will be encouraged to finish it safely as soon as possible. A shorter time indicates better function.
Change of 15-m walk test | The day before operation day, and 1, 3, 6 months after surgery
  Gait speed shows good reliability and is valid to assess physical mobility. A 15-mile straight line will be mounted on a flat surface. The patient will be required to walk down the line at the maximal speed. He/She will be encouraged to finish it safely as soon as possible. A shorter time indicates better function.

SECONDARY OUTCOMES:
Length of hospitalization | The duration between admission and discharge
Narcotic use during hospitalization | The duration between admission and discharge
Return-to-work status | up to 6 months after surgery
Adverse events | up to 6 months after surgery
  The rate of infection and the rate of re-operation (including: dural tear, cage migration and retropulsion, and screw loosening).

CONTACTS AND LOCATIONS:
Overall Officials: Heng-Wei Liu, Doctor, Study Chair — ShuangHo Hospital
Locations (1):
- Taipei Medical University-Shuang Ho Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No